CLINICAL TRIAL: NCT03518255
Title: e-Natureza: Affective Validation of Nature Images as a Complementary Resource for Promoting Well-being in Hospital Environment
Brief Title: e-Natureza Project - Affective Validation of Nature Images for Hospital Use
Acronym: E-natureza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: e-Natureza
Record Dates: First submitted 2018-03-12; First posted 2018-05-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cancer
Keywords: Nursing Care; Complementary therapies; Oncological Nursing; Photography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Masking Description: This study has no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This control group will not receive an intervention.
- Nature video (Experimental): A pre-validated nature images video will be shown to the patient during their chemotherapy session. After thirty minutes of the start of the chemotherapy session, the patient you will receive a notebook (specific to the study and blocked for other functions) that he can watch a presentation of nature images. It will be four videos with fifteen minutes each one.
  Interventions: Other: Nature video

INTERVENTIONS:
Other: Nature video — After signing the Informed Consent Form, the participants will respond to a demographic questionnaire to characterize the sample and then they will watch nature videos. After that, will be applied a scale questionnaire about the physical and psychological symptoms of chemotherapy in the positive and negative mood of that patient.
  Arms: Nature video

SUMMARY:
Randomized clinical trial about the evaluation of the use of nature photographs in the positive and negative affects of oncological patients.

DETAILED DESCRIPTION:
In recent decades there has been growing interest from researchers in understanding how the adoption of natural elements in daily life, even in hospitals, can characterize restorative environments and reflect in better health for patients. Contact with nature can be done indirectly through photographs. This clinical trial aims to verify the therapeutic potential of the nature images, previously validated in another part of this study, in the care of cancer patients undergoing chemotherapy. Anchored on the assumptions of the theory of Biophilia, and the environmental theory of Florence Nightingale our study hypothesis is that this intervention promotes well-being and promote more positive mood states, and reduce symptoms resulting from the treatment during chemotherapy session.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation;
* Signed in the Informed Consent Form;
* Who are undergoing chemotherapy treatment;
* Patients need to be on the first chemotherapy session, independently of oncological disease;
* Patients with clinical conditions and preserved communication function, in other words, lucid patients.

Exclusion Criteria:

* Blind patients;
* Patients without the capacity for judgment, in other words, with dementia;
* Patients who have their clinical condition aggravated during the chemotherapy session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | Change from Baseline positive and negative affects at immediate post intervention, through study completion, an average of 1 year
  The questionnaire aims to verify the positive and negative affects of participants in oncologic treatment before and after their first chemotherapy session, in order to verify if after the intervention, the negative affects decrease and the positive ones increase. Each questionnaire will be analyzed individually.

SECONDARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS-Br) | Change from Baseline Edmonton Symptoms at immediate post intervention, through study completion, an average of 1 year
  This tool is designed to assist in the assessment of nine symptoms common in cancer patients: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing and shortness of breath, (there is also a line labelled "Other Problem"). The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity. It does not have final classification scores. It measures the frequency and intensity of symptoms presented at the time of its application.

OTHER OUTCOMES:
The Connectedness to Nature Scale | Single baseline measurement
  The Nature Connection Scale is used to verify the affective aspect of the person-environment relationship. It is composed of 14 items, which are answered in a scale of 5 points, ranging from 1 (I totally disagree) to 5 (I totally agree). The higher the score, the greater the individual's connection with nature.
Nature Relatedness Questionnaire | Single baseline measurement
  The 21-item Nature Relatedness Scale (NR) assesses subjective connectedness with the natural environment. Participants respond to statements using a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree) and items are averaged with higher scores indicating stronger connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein- Research Institute; Gustavo B Borba, PhD, Study Chair — Federal Technological University of Paraná; João M Rosa, BAA, Study Chair — National Geografic; Elivane S Victor, BSS, Study Chair — Hospital Israelita Albert Einstein- Research Institute; Daniela R Dal Fabbro, BSN, Study Chair — Hospital Israelita Albert Einstein- Research Institute; Giulia C Lima, BSN, Study Chair — Hospital Israelita Albert Einstein- Research Institute; Tinely B Souza, Student, Study Chair — Hospital Israelita Albert Einstein- Research Institute; Fábio S Romano, BSc, Study Chair — Hospital Israelita Albert Einstein- Oncological Unit; Erika H Zaher, PhD, Study Chair — Butanta Institute; Luciano M Lima, MSc, Study Chair — Butanta Institute
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leao ER, Dal Fabbro DR, Oliveira RB, Santos IR, Victor ED, Aquarone RL, Andrade CB, Ribeiro VF, Oliveira RC, Friedlander R, Ferreira DS. Stress, self-esteem and well-being among female health professionals: A randomized clinical trial on the impact of a self-care intervention mediated by the senses. PLoS One. 2017 Feb 27;12(2):e0172455. doi: 10.1371/journal.pone.0172455. eCollection 2017. PMID 28241070

DOCUMENTS (2):
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT03518255/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT03518255/Prot_SAP_001.pdf